CLINICAL TRIAL: NCT05989932
Title: Esperienza Real-world Sull'Uso di Upadacitinib Nel Trattamento Della Dermatite Atopica Moderata-severa Dell'Adulto
Brief Title: Real-world Experience on the Use of Upadacitinib in the Treatment of Moderate-severe Adult Atopic Dermatitis (ERUDA)
Acronym: ERUDA
Status: Completed | Type: Observational
Sponsor: Societa Italiana di Dermatologia Medica, Chirurgica, Estetica e di Malattie Sessualmente Trasmesse (Other)
Responsible Party: Sponsor
Other Study IDs: SID02
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Upadacitinib — Real-world on the use of Upadacitinib

SUMMARY:
Real-world experience on the use of Upadacitinib in the treatment of Adult moderate-severe atopic dermatitis

DETAILED DESCRIPTION:
Atopic dermatitis (DA) is a chronic-recurrent inflammatory skin disease with high prevalence in children. Clinical remission is frequently observed during or after childhood although it may persist and/or recur, even after long and transient remission, in adulthood. In addition, in some patients the DA begins in adulthood: in these cases, we speak of DA adult-onset. In addition to the diagnostic framework, it is also important in clinical practice to assess the severity of the disease on which the choice of treatment is based, which will also take into account other factors such as: possible comorbidities, Previously performed therapies and patient needs. For the management of moderate-severe forms of atopic dermatitis topical drugs, phototherapy, traditional immunomodulating drugs and a biological drug are currently available. Compared to other chronic inflammatory skin diseases the therapeutic paraphernalia should be considered limited, with most systemic drugs that have no indication for the treatment of DA (off-label use).

In the pipeline there are numerous drugs that have reached an advanced stage of development. These include upadacitinib, a new-generation oral drug (small molecule) that selectively inhibits the signal mediated by Janus kinases 1 (JAK-1), has recently received approval for treatment of DA by EMA and AIFA to begin compassionate use of patients deemed contraindicated, intolerant, and/or non-responsive to traditional systemic therapies and biological therapy.

* Evaluation of the effectiveness of upadacitinib using the EASI score Secondary objectives
* Evaluation of the safety profile of upadacitinib
* Predictive factors of treatment response
* Assessment of patient quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years
2. Signature of informed consent
3. Diagnosis of moderate and/or severe DA by a dermatologist specialist
4. Approval of the compassionate use of upadacitinib

Exclusion Criteria:

1. Patient unable to give informed consent prior to any collection procedure study data
2. unable to complete the procedures required for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The nature of the study is descriptive. Each center is committed to enlist consecutively all adult patients diagnosed with moderate-severe atopic dermatitis treated with upadacitinib
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Dermatology life quality index (DLQI) | from enrollment up to 48 weeks
  Assessment of the patient's quality of life. There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life) --> 0-1 = No effect on patient's life, 2-5 = Small effect, 6-10 = Moderate effect, 11-20 = Very large effect, 21-30 = Extremely large effect
Patient-oriented eczema measure (POEM) | From enrollment up to 48 weeks
  The Patient Oriented Eczema Measure (POEM) is a simple, validated self-report questionnaire used for monitoring atopic eczema severity. It records seven symptoms shown to be important to patients, like itchy, sleep, bleeding ect.. Each of the seven questions carries equal weight and is scored from 0 to 4 as follows: No days = 0; 1-2 days = 1; 3-4 days = 2; 5-6 days = 3; Every day = 4. The meaning is: 0 to 2 = Clear or almost clear; 3 to 7 = Mild eczema; 8 to 16 = Moderate eczema; 17 to 24 = Severe eczema; 25 to 28 = Very severe eczema.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Fondazione Policlinico Gemelli, Roma, ROMA, Italy

IPD SHARING:
Plan to Share IPD: Undecided